CLINICAL TRIAL: NCT06966037
Title: Evaluation of Uric Acid Levels in Pediatric Patients With Migraine
Brief Title: Uric Acid Levels and Migraine in Children
Status: Completed | Type: Observational
Sponsor: Aysen Orman (Other)
Responsible Party: Sponsor-Investigator, Aysen Orman, Mersin University, Mersin University
Organization: Mersin University (Other)
Other Study IDs: Balikesir University
Record Dates: First submitted 2025-04-24; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Migraine in Children
Keywords: migraine; children; uric acid levels
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Comparison of Laboratory Parameters Between Groups: The present study aims to compare serum uric acid levels between pediatric patients with migraine and a control group

SUMMARY:
Migraine is recognized as one of the most prevalent neurological disorders. The exact pathophysiological mechanisms underlying migraine have not yet been fully elucidated. The present study aims to compare serum uric acid levels between pediatric patients with migraine and a control group. Additionally, this study seeks to explore the potential relationship between migraine attack frequency and gender differences in pediatric patients

DETAILED DESCRIPTION:
Migraine is recognized as one of the most prevalent neurological disorders. The exact pathophysiological mechanisms underlying migraine have not yet been fully elucidated. The present study aims to compare serum uric acid levels between pediatric patients with migraine and a control group. Additionally, this study seeks to explore the potential relationship between migraine attack frequency and gender differences in pediatric patients Patients diagnosed with migraine were included as the study group, while the control group consisted of patients who presented to the pediatric neurology clinic during the same period for neuromotor development follow-up examinations.

Migraine patients are influenced by multiple factors, including dietary habits, levels of physical activity, and various psychosocial determinants.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with migraine

Exclusion Criteria:

Cerebral palsy Non-migraine headache Epilepsy Multiple congenital anomalies Congenital metabolic diseases Control group

Inclusion Criteria:

Healthy children Exclusion Criteria Neuromotor developmental delay Multiple congenital anomalies Non-migraine headache Epilepsy

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients diagnosed with migraine were included as the study group, while the control group consisted of patients who presented to the pediatric neurology clinic during the same period for neuromotor development follow-up examinations.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of Uric Acid Levels in Pediatric Patients with Migraine | 01.08.2019 and 01.03.2024
  Migraine represents a significant neurological condition affecting individuals across all age groups, with a reported prevalence of 7.7% among children and adolescents. According to the widely accepted neurogenic inflammation hypothesis, sterile inflammation occurs in the dura mater surrounding the brain as a result of neuropeptide release from perivascular trigeminal nerve endings, leading to sensitization of sensory neurons .Uric acid is known to function as a potent endogenous antioxidant and free radical scavenger within the human body. It has been suggested that uric acid exerts dual effects on the central nervous system, demonstrating both neuroprotective and neurotoxic properties depending on its concentration. Although uric acid may enhance antioxidant and anti-inflammatory responses at physiological concentrations, it has been suggested that excessively elevated serum uric acid levels may contribute to increased oxidative stress and subsequent neuronal damage. The primary ou

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol